CLINICAL TRIAL: NCT01748721
Title: Study of the TEM-1 Antibody, MORAb-004 (IND# 103821), in Children With Recurrent or Refractory Solid Tumors
Brief Title: MORAb-004 in Treating Young Patients With Recurrent or Refractory Solid Tumors or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Morphotek (Industry)
Collaborators: National Cancer Institute (NCI) (NIH); Children's Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADVL1213; NCI-2012-01702 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); U01CA097452 (NIH)
Record Dates: First submitted 2012-12-11; First posted 2012-12-12 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2015-12

CONDITIONS: Adult Nasal Type Extranodal NK/T-cell Lymphoma; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Childhood Burkitt Lymphoma; Childhood Diffuse Large Cell Lymphoma; Childhood Immunoblastic Large Cell Lymphoma; Childhood Nasal Type Extranodal NK/T-cell Lymphoma; Cutaneous B-cell Non-Hodgkin Lymphoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Hepatosplenic T-cell Lymphoma; Intraocular Lymphoma; Nodal Marginal Zone B-cell Lymphoma; Noncutaneous Extranodal Lymphoma; Peripheral T-cell Lymphoma; Post-transplant Lymphoproliferative Disorder; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Childhood Anaplastic Large Cell Lymphoma; Recurrent Childhood Grade III Lymphomatoid Granulomatosis; Recurrent Childhood Large Cell Lymphoma; Recurrent Childhood Lymphoblastic Lymphoma; Recurrent Childhood Small Noncleaved Cell Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Small Lymphocytic Lymphoma; Recurrent/Refractory Childhood Hodgkin Lymphoma; Refractory Hairy Cell Leukemia; Small Intestine Lymphoma; Splenic Marginal Zone Lymphoma; T-cell Large Granular Lymphocyte Leukemia; Testicular Lymphoma; Unspecified Adult Solid Tumor, Protocol Specific; Unspecified Childhood Solid Tumor, Protocol Specific; Waldenström Macroglobulinemia
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Intraocular Lymphoma; Lymphoma, B-Cell, Marginal Zone; Lymphoma, T-Cell, Peripheral; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence; Leukemia, Hairy Cell; Leukemia, Large Granular Lymphocytic; Waldenstrom Macroglobulinemia | interventions — ontuxizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (MORAb-004) (Experimental): Patients receive anti-endosialin/TEM1 monoclonal antibody MORAb-004 IV on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 13 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: anti-endosialin/TEM1 monoclonal antibody MORAb-004; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: anti-endosialin/TEM1 monoclonal antibody MORAb-004 — Given IV
  Other Names: MORAb-004
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Optional correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of MORAb-004 in treating young patients with recurrent or refractory solid tumors or lymphoma. Monoclonal antibodies, such as MORAb-004, can block cancer growth in different ways. Some block the ability of cancer to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the maximum tolerated dose (MTD) and/or recommended phase 2 dose of MORAb-004 (anti-endosialin/TEM1 monoclonal antibody MORAb-004) administered as an intravenous infusion every week to children with refractory solid tumors.

II. To define and describe the toxicities of MORAb-004 administered on this schedule.

III. To characterize the pharmacokinetics of MORAb-004 in children with refractory cancer.

IV. To monitor for the development of human anti-human antibody (HAHA) in children receiving MORAb-004.

SECONDARY OBJECTIVES:

I. To preliminarily define the antitumor activity of MORAb-004 within the confines of a phase 1 study.

II. To examine tumor endothelial marker-1 (TEM-1) and PDGFRB levels in tissue and plasma samples as potential biomarkers of MORAb-004 activity.

III. To correlate baseline expression of TEM-1 and PDGFRB (in issue and plasma)with clinical parameters including disease response in an exploratory manner.

OUTLINE: This is a dose escalation study.

Patients receive anti-endosialin/TEM1 monoclonal antibody MORAb-004 intravenously (IV) on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 13 courses in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsed or refractory solid tumors or lymphoma, excluding central nervous system (CNS) tumors, are eligible; patients must have had histologic verification of malignancy at original diagnosis or relapse; (patients with primary CNS tumors, known CNS metastases, or a prior history of CNS metastases are not eligible)
* Patients must have either measurable or evaluable disease
* Patient's current disease state must be one for which there is no known curative therapy or therapy proven to prolong survival with an acceptable quality of life
* Karnofsky >= 50% for patients > 16 years of age and Lansky >= 50 for patients =< 16 years of age; Note: patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Patients must have fully recovered from the acute toxic effects of all prior anti-cancer chemotherapy
* At least 21 days after the last dose of myelosuppressive chemotherapy (42 days if prior nitrosourea)
* At least 14 days after the last dose of a long-acting growth factor (e.g. Neulasta) or 7 days for short-acting growth factor; for agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur; the duration of this interval must be discussed with the study chair
* At least 7 days after the last dose of a biologic agent; for agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur; the duration of this interval must be discussed with the study chair
* At least 42 days after the completion of any type of immunotherapy, e.g. tumor vaccines
* At least 3 half-lives of the antibody after the last dose of a monoclonal antibody
* At least 14 days after local palliative radiotherapy (XRT) (small port); at least 150 days must have elapsed if prior total-body irradiation (TBI), craniospinal XRT or if >= 50% radiation of pelvis; at least 42 days must have elapsed if other substantial bone marrow (BM) radiation
* No evidence of active graft vs. host disease and at least 56 days must have elapsed after transplant or stem cell infusion
* For patients with solid tumors without known bone marrow involvement:
* Peripheral absolute neutrophil count (ANC) >= 1000/mm^3
* Platelet count >= 100,000/mm^3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment)
* For patients with known bone marrow metastatic disease:
* ANC >= 750/mm^3
* Platelet count >= 75,000/mm^3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment)
* Patients with known bone marrow metastatic disease will not be evaluable for hematologic toxicity; these patients must not be known to be refractory to red cell or platelet transfusion; at least 5 of every cohort of 6 patients with a solid tumor or lymphoma must be evaluable for hematologic toxicity; if dose-limiting hematologic toxicity is observed, all subsequent patients enrolled must be evaluable for hematologic toxicity
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70ml/min/1.73 m^2 OR a serum creatinine based on age/gender as follows:

  * =< 0.6 mg/dL for patients age 1 to < 2 years
  * =< 0.8 mg/dL for patients age 2 to < 6 years
  * =< 1 mg/dL for patients age 6 to 10 2 years
  * =< 1.2 mg/dL for patients age 10 to < 13 years
  * =< 1.4 mg/dL for female patients age >= 13 years
  * =< 1.5 mg/dL for male patients age 13 to < 16 years
  * =< 1.7 mg/dL for male patients age >= 16 years
* Bilirubin (sum of conjugated + unconjugated) =< 1.5 x upper limit of normal (ULN) for age
* Serum glutamic pyruvic transaminase (SGPT) (alanine aminotransferase [ALT]) =< 110 U/L; for the purpose of this study, the ULN for SGPT is 45 U/L
* Serum albumin >= 2 g/dL
* Activated partial thromboplastin time (aPTT) and prothrombin time (PT) =< 1.5 x ULN
* All patients and/or their parents or legally authorized representatives must sign a written informed consent; assent, when appropriate, will be obtained according to institutional guidelines
* Tissue blocks or slides must be sent per Section 8.5. If tissue blocks or slides are unavailable, the study chair must be notified prior to enrollment.

Exclusion Criteria:

* Pregnant or breast-feeding women will not be entered on this study; pregnancy tests must be obtained in girls who are post-menarchal; males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method
* Patients receiving chronic systemic corticosteroids are not eligible
* Patients who are currently receiving another investigation drug are not eligible
* Patients who are currently receiving other anti-cancer agents are not eligible
* Patients who are receiving cyclosporine, tacrolimus or other agents to prevent graft-versus-host disease post bone marrow transplant are not eligible for this trial
* Patients who have known human immunodeficiency virus (HIV), viral hepatitis, or an uncontrolled infection are not eligible
* Patients with primary CNS tumors are excluded
* Patients with prior history of or known metastatic CNS disease involvement are excluded; (Note: CNS imaging for patients without a known history of CNS disease is only required if clinically indicated)
* Patients who have had or are planning to have the following invasive procedures are not eligible:

  * Major surgical procedure, laparoscopic procedure, open biopsy or significant traumatic injury within 28 days prior to enrollment
  * Central line placement or subcutaneous port placement is not considered major surgery but must be placed at least 3 days prior to enrollment for external lines (e.g. Hickman or Broviac) and at least 7 days prior to enrollment for subcutaneous port
  * Core biopsy within 7 days prior to enrollment
  * Fine needle aspirate within 7 days prior to enrollment
* Patients who have received prior solid organ transplantation are not eligible
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible
* Patients with history of clinically significant bleeding risk (including evidence of active bleeding: intratumoral hemorrhage by current imaging, or bleeding diathesis; bleeding/coagulation disorder; active fracture; non-healing wound; and active gastric ulcer) are not eligible

Ages: 13 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 27 (Actual)
Dates: Start 2013-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
MTD, defined as the maximum dose at which fewer than one-third of patients experience dose-limiting toxicities (DLT) graded according to the revised National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | Up to 4 weeks
Incidence of toxicities, graded according to NCI CTCAE version 4.0 | Up to 3 years
  A descriptive summary of all toxicities will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Robin Norris, Principal Investigator — Children's Oncology Group
Locations (20):
- United States (20):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Children's Hospital of Orange County, Orange, California
  - University of California San Francisco Medical Center - Parnassus, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta-Egleston, Atlanta, Georgia
  - Ann and Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - University of Minnesota Cancer Center-Fairview, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies & Children's Hospital, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Norris RE, Fox E, Reid JM, Ralya A, Liu XW, Minard C, Weigel BJ. Phase 1 trial of ontuxizumab (MORAb-004) in children with relapsed or refractory solid tumors: A report from the Children's Oncology Group Phase 1 Pilot Consortium (ADVL1213). Pediatr Blood Cancer. 2018 May;65(5):e26944. doi: 10.1002/pbc.26944. Epub 2018 Jan 2. PMID 29292843